## Revitalize Cognition: Near Infrared Stimulation in Older Adults NCT06688357

11/13/2024

Updated Statistical Plan

## **Updated Statistical Analysis Plan**

Due to the small N, we examined cognitive and emotion outcome variables using change scores (post intervention – baseline). These change scores were evaluated as a function of treatment group (active, sham) using independent t-tests. Cohen's D effect sizes were computed to guide selection of potential cognitive measures for use in future clinical trials, as appropriate.